CLINICAL TRIAL: NCT03457870
Title: Investigating the Impact of Intermittent Energy Restriction and Chewing on Neural Stem Cell Ageing and Adult Hippocampal Neurogenesis: The ChANgE Study
Brief Title: Intermittent Energy Restriction and Chewing on Neural Stem Cell Ageing and Adult Hippocampal Neurogenesis Associated Cognition
Acronym: ChANgE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: Medical Research Council (Other Government); Mars, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Change 2018
Record Dates: First submitted 2018-02-23; First posted 2018-03-08 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Aging; Cognitive Decline
Keywords: Intermittent fasting; Adult hippocampal neurogenesis; Mastication; Pattern separation; Recognition memory; Klotho
MeSH Terms: conditions — Cognitive Dysfunction; Intermittent Fasting | interventions — Mastication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Intermittent Energy Restriction (Experimental): Dietary intervention: Intermittent energy restriction
  Interventions: Behavioral: Intermittent Energy Restriction
- Chewing (Experimental): Mastication intervention: chewing
  Interventions: Behavioral: Chewing
- Chewing + Intermittent Energy Restriction (Experimental): Dietary and mastication intervention: Intermittent energy restriction and chewing
  Interventions: Behavioral: Chewing + Intermittent Energy Restriction
- Control (No Intervention): No intervention: Control

INTERVENTIONS:
Behavioral: Intermittent Energy Restriction — Dietary advice to follow a 5:2 diet.
  Arms: Intermittent Energy Restriction
Behavioral: Chewing — Asked to chew 1 piece of gum for 10 minutes 3 times a day.
  Arms: Chewing
Behavioral: Chewing + Intermittent Energy Restriction — Dietary advice to follow a 5:2 diet. Asked to chew 1 piece of gum for 10 minutes 3 times a day.
  Arms: Chewing + Intermittent Energy Restriction

SUMMARY:
Extended bouts of periodic mastication and intermittent energy restriction (IER) may improve cognitive performance in the context of adult hippocampal neurogenesis in an ageing population. A randomised controlled parallel design trial will determine the impact of a 3 month IER diet (2 consecutive days of very low calorie diet and 5 days of normal eating) and a mastication intervention (1 piece of gum chewed for 10 minutes 3 times a day) in comparison to a control on neurogenesis-associated cognitive measures and circulating levels of the anti-ageing protein Klotho.

DETAILED DESCRIPTION:
Nutrition and human health are strongly related. Altering overabundance through fasting/calorie-restricted diets has profound effects on homeostasis, tissue regeneration, and cancer. Tissue stem cells respond to the physiological changes that occur during fasting through dynamic shifts in their metabolism. Restricting energy intake in mice or introducing mutations in nutrient-sensing pathways can extend lifespans by as much as 50%. Post-mortems reveal that tumours, heart problems, neurodegeneration and metabolic disease are generally reduced/delayed in long-lived mice. Therefore, extending lifespan by energy restriction (ER) also seems to increase 'healthspan', the time lived without chronic age-related conditions. These insights have hardly made a dent in human medicine. Molecular and cellular insights should be established in humans to validate interventions such as ER to delay ageing and associated conditions e.g. cognitive decline (Murphy et al., 2014).

Stem cells from the central nervous system also respond to ER. Recently, the Thuret lab have found that ER, in the absence of malnutrition, promotes hippocampal stem cells to proliferate and differentiate into new-born neurons. Because these new postnatal hippocampal neurons have been shown to play a role in cognition, ER also promoted enhanced cognition in rodents (Zainuddin et al., 2012; de Lucia et al., 2017; Thuret et al., 2012). This phenomenon of neurogenesis, the process by which new neurons are generated from neural stem cells, is also occurring in humans (Spalding et al., 2013). It is a tightly regulated process occurring in the mammalian hippocampus which is an environmentally responsive brain structure known to regulate learning, memory and mood. Proposed functions of adult hippocampal neurogenesis (AHN). include enhancing recognition memory, the ability to recognise previously encountered stimuli, and pattern separation, the ability to differentially encode small changes in similar inputs (Clelland et alk., 2009; Sahay et al., 2011). It has been posited that calorie restriction may increase neurogenesis as a "cellular relic" of intermittent feeding patterns during evolution as a response to alternating periods of famine and abundant food (Murphy & Thuret, 2015). Human trials have found significant improvements in verbal recognition memory after 30% reduction in calorie intake (Witte et al., 2009). Also, intermittent fasting in humans has been associated with significant increases in brain activation volume in areas involved in brain function control and plasticity(Belaïch et al., 2016). Food texture and mastication have also been implicated in AHN and cognitive ability (Smith et al., 2016). Decreased mastication due to the removal of molars and edentulism in both humans and animals have a negative impact on AHN and associated cognition. Human populations, in particular, have shown a close association between masticatory function, cognitive status and age-related neurodegeneration in the elderly (Miura et al., 2003). The exact mechanism by which mastication affects cognition is unknown.

Research question: In older, overweight participants does IER and/or extended periods of mastication enhance performance inhippocampus-dependent memory tasks and increase anti-ageing marker Klotho?

Objectives:

1. A randomised controlled parallel-design trial will determine the impact of an IER diet (2 consecutive days of a very low calorie diet, 5 days of normal healthy eating for 3 months) and/or extended periods of mastication (10 minutes 3 times a day for 3 months) compared to a control group (continued habitual eating behaviour, dietary patterns) on primary outcome variables (MST and Klotho) in older, healthy participants with overweight or class I obesity.
2. To assess the impact of an IER diet and extended periods of mastication on secondary outcomes variables including body composition, mood and sleep.
3. To explore whether extended periods of mastication can be utilised as a weight loss/fasting aid.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects.
* 60+ years of age at the time of consent.
* BMI 25-35.

Exclusion Criteria:

* Subject is unable to understand the participant information sheet.
* Subject is unable to understand and/or completely perform the cognitive testing.
* Chews more than 3 sticks of gum per month, including nicotine replacement gum.
* Unable to provide written informed consent.
* Impaired vision that is not corrected.
* Does not agree to maintain their habitual exercise routine.
* Is not in general good health on the basis of medical history.
* Unwilling to chew gum for 3 times a day for 12 weeks.
* Unwilling to maintain an intermittent fasting diet regime.
* Unwilling to have blood taken.
* History of or are currently diagnosed with a significant psychiatric disorder (e.g. schizophrenia, anxiety, PTSD).
* Subject has any neurological disorder that could produce cognitive deterioration (e.g. Alzheimer's disease, Parkinson's disease, stroke).
* History of traumatic brain injury, stroke or any other medical conditions causing cognitive impairment.
* Has uncontrolled epilepsy or is prone to fainting.
* Participated in a weight management drug trial in previous 3 months.
* Has undergone bariatric surgery.
* Known or suspected of alcohol abuse defined as >14 drinks per week (1 drink = 1 pint of beer, 1 large glass of wine or 50ml spirit).
* Gastrointestinal or liver disease.
* Subject has a sleep disorder or an occupation where sleep during the overnight hours is irregular.
* Subjects taking the following prescription medications: Donepezil (Aricept), Galantamine (Reminyl), Rivastigmine (Exelon), Tacrine (Cognex), Bethanechol (Urecholine), Memantine (Namenda) Selegiline (Eldepryl) or any other medication for cognitive impairment.
* Subject has a known sensitivity to the study product.
* Individual has a condition the chief investigator believes would interfere with his or her ability to provide informed consent, comply with the study protocol, might confound the interpretation of study results or put the subject at undue risk.

Min Age: 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2018-04-18 (Actual); Primary Completion 2020-03-23 (Actual); Study Completion 2020-03-23 (Actual)

PRIMARY OUTCOMES:
Serum Klotho concentration | Baseline
  Anti-ageing longevity protein
Serum Klotho concentration | Day 42
  Anti-ageing longevity protein
Serum Klotho concentration | Day 84
  Anti-ageing longevity protein
Mnemonic Similarity Task | Baseline
  Neurogenesis-associated cognition
Mnemonic Similarity Task | Day 42
  Neurogenesis-associated cognition

SECONDARY OUTCOMES:
Body weight | Baseline
Body weight | Day 42
Body weight | Day 84
Body fat percentage | Baseline
Body fat percentage | Day 42
Body fat percentage | Day 84
Body Mass Index | Baseline
Body Mass Index | Day 42
Body Mass Index | Day 84
Waist circumference | Baseline
Waist circumference | Day 42
Waist circumference | Day 84
Hip circumference | Baseline
Hip circumference | Day 42
Hip circumference | Day 84
Patient Health Questionnaire | Baseline
  Questionnaire
Patient Health Questionnaire | Day 42
  Questionnaire
Patient Health Questionnaire | Day 84
  Questionnaire
Zung Self-Rating Anxiety Scale | Baseline
  Questionnaire - Scale can be scored from 20 (normal) to 80 (extreme anxiety levels). The total score is reported.
Zung Self-Rating Anxiety Scale | Day 42
  Questionnaire
Zung Self-Rating Anxiety Scale | Day 84
  Questionnaire
Pittsburgh Sleep Quality Index | Baseline
  Questionnaire
Pittsburgh Sleep Quality Index | Day 42
  Questionnaire
Pittsburgh Sleep Quality Index | Day 84
  Questionnaire
Plasma glucose concentration | Baseline
  Fasting
Plasma glucose concentration | Day 42
  Fasting
Plasma glucose concentration | Day 84
  Fasting
Cholesterol | Baseline
  Fasting
Cholesterol | Day 42
  Fasting
Cholesterol | Day 84
  Fasting
Triglycerides | Baseline
  Fasting
Triglycerides | Day 42
  Fasting
Triglycerides | Day 84
  Fasting
High Density Lipoprotein | Baseline
  Fasting
High Density Lipoprotein | Day 42
  Fasting
High Density Lipoprotein | Day 84
  Fasting
Low Density Lipoprotein | Baseline
  Fasting
Low Density Lipoprotein | Day 42
  Fasting
Low Density Lipoprotein | Day 84
  Fasting
Total/HDL Cholesterol Ratio | Baseline
  Fasting
Total/HDL Cholesterol Ratio | Day 42
  Fasting
Total/HDL Cholesterol Ratio | Day 84
  Fasting
Plasma adiponectin concentration | Baseline
  Fasting
Plasma adiponectin concentration | Day 42
  Fasting
Plasma adiponectin concentration | Day 84
  Fasting
Plasma leptin concentration | Baseline
  Fasting
Plasma leptin concentration | Day 42
  Fasting
Plasma leptin concentration | Day 84
  Fasting
Plasma beta-hydroxybutrate concentration | Baseline
  Fasting
Plasma beta-hydroxybutrate concentration | Day 42
  Fasting
Plasma beta-hydroxybutrate concentration | Day 84
  Fasting
Plasma total cholesterol concentration | Baseline
  Fasting
Plasma total cholesterol concentration | Day 42
  Fasting
Plasma total cholesterol concentration | Day 84
  Fasting
Plasma low density lipoprotein (LDL) cholesterol concentration | Baseline
  Fasting
Plasma LDL cholesterol concentration | Day 42
  Fasting
Plasma LDL cholesterol concentration | Day 84
  Fasting
Plasma high density lipoprotein (HDL) cholesterol concentration | Baseline
  Fasting
Plasma HDL cholesterol concentration | Day 42
  Fasting
Plasma HDL cholesterol concentration | Day 84
  Fasting
Plasma triglyceride concentration | Baseline
  Fasting
Plasma triglyceride concentration | Day 42
  Fasting
Plasma triglyceride concentration | Day 84
  Fasting
Plasma total cholesterol:HDL cholesterol ratio | Baseline
  Fasting
Plasma total cholesterol:HDL cholesterol ratio | Day 42
  Fasting
Plasma total cholesterol:HDL cholesterol ratio | Day 84
  Fasting

OTHER OUTCOMES:
Adverse events | Baseline until endpoint: Day 84

CONTACTS AND LOCATIONS:
Overall Officials: Sandrine Thuret, PhD, Principal Investigator — King's College London; Wendy L Hall, PhD, Principal Investigator — King's College London
Locations (1):
- Diabetes & Nutritional Sciences Division, King's College London, Franklin-Wilkins Building, 150 Stamford St, London, England, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Murphy T, Dias GP, Thuret S. Effects of diet on brain plasticity in animal and human studies: mind the gap. Neural Plast. 2014;2014:563160. doi: 10.1155/2014/563160. Epub 2014 May 12. PMID 24900924
- [Background] Witte AV, Fobker M, Gellner R, Knecht S, Floel A. Caloric restriction improves memory in elderly humans. Proc Natl Acad Sci U S A. 2009 Jan 27;106(4):1255-60. doi: 10.1073/pnas.0808587106. Epub 2009 Jan 26. PMID 19171901
- [Background] Akazawa Y, Kitamura T, Fujihara Y, Yoshimura Y, Mitome M, Hasegawa T. Forced mastication increases survival of adult neural stem cells in the hippocampal dentate gyrus. Int J Mol Med. 2013 Feb;31(2):307-14. doi: 10.3892/ijmm.2012.1217. Epub 2012 Dec 18. PMID 23254518
- [Background] Smith, N., Miquel-Kergoat, S. & Thuret, S., 2016. The impact of mastication on cognition: Evidence for intervention and the role of adult hippocampal neurogenesis. Nutrition and Aging, 3(2-4), pp.115-123